CLINICAL TRIAL: NCT01212926
Title: Early Detection of Anthracycline Cardiotoxicity by Echocardiographic Analysis of Myocardial Deformation in 2D Strain
Acronym: CA2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2009/23
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Leukemia; Cardiac Toxicity
MeSH Terms: conditions — Leukemia; Cardiotoxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- analysis of myocardial deformation in 2D strain (Experimental)
  Interventions: Device: Echographic analysis of myocardial deformation in 2D strain

INTERVENTIONS:
Device: Echographic analysis of myocardial deformation in 2D strain

SUMMARY:
It is now accepted that the anticancer properties of anthracyclines were allowed in many malignancies improve the prognosis of affected populations.

However, the cardiotoxicity of anthracyclines is responsible for an interruption of this treatment by alteration of potentially irreversible myocardial contraction and high mortality.

An earlier detection of adverse myocardial anthracycline chemotherapy would allow the adaptation of the regimen by reducing the number of interruptions of antitumor and strengthening monitoring. Optimizing the therapeutic antitumor and generate an increase in survival of patients treated.

DETAILED DESCRIPTION:
Analysis of myocardial deformation in its longitudinal component, circumferential and radial, is a new echocardiographic technique for evaluating myocardial function, which has demonstrated its superiority compared to LVEF in many clinical situations. It therefore seems promising to evaluate this new tool in the earlier detection of adverse myocardial chemotherapy with anthracyclines. The ultimate goal is indeed to determine a reliable and reproducible parameter for cardiac toxicity diagnostic to avoid chemotherapy interruption, thus improving the survival of these patients.

The main objective of this project is to evaluate the association between changes in myocardial deformation longitudinal 2D strain echocardiography between baseline and 6 weeks after initiation of anthracycline therapy for acute leukemia and the occurrence of impaired left ventricular function within 12 months after starting treatment.

It is a prognostic study of clinical-looking, without randomization. The inclusion will take place over a period of 12 months with a total follow-up of 12 months.

The analysis will focus on the identification of parameters predictive of alteration of Fe VG.

ELIGIBILITY:
Inclusion Criteria:

* Patient female or male aged between 18 and 65
* Patients with a haematological disease and ran for a first-line chemotherapy including anthracycline
* Patients with a predict cardiovascular score to 10 years below 20% or if higher, with a stress echocardiography using dobutamine, negative, for less than six months.
* Patient or affiliate receiving social security
* Patient informed consent and having oral and written

Exclusion Criteria:

* A history of chemotherapy or radiotherapy of the left hemithorax
* Significant coronary artery disease: a history of angioplasty, stent, CABG, predict cardiovascular score to 10 years over 20% of stress echocardiography and dobutamine positive (three positive segments)
* Left ventricular hypertrophy (diastolic septum ≥ 10 mm and diastolic posterior wall ≥ 10 mm)
* One or more significant valvulopathy: Rao, RM medium or tight, IM, IT and CAI ≥ grade 2
* Secondary or primary cardiomyopathy (LVEF ≤ 50%)
* Pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-09-28 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2015-05-25 (Actual)

PRIMARY OUTCOMES:
determination of longitudinal myocardial deformation by echography with 2D strain analysis after 6 weeks of anthracycline chemotherapy. | 6 weeks
determination of longitudinal myocardial deformation by echography with 2D strain analysis after 3 months of anthracycline chemotherapy. | 3 months
determination of longitudinal myocardial deformation by echography with 2D strain analysis after 6 months of anthracycline chemotherapy. | 6 months
determination of longitudinal myocardial deformation by echography with 2D strain analysis after 9 months of anthracycline chemotherapy. | 9 months
determination of longitudinal myocardial deformation by echography with 2D strain analysis after 12 months of anthracycline chemotherapy. | 12 months

SECONDARY OUTCOMES:
determination of radial and circumferential myocardial deformation by echography with 2D strain analysis after 6 weeks of anthracycline chemotherapy. | 6 weeks
determination of radial and circumferential myocardial deformation by echography with 2D strain analysis after 3 months of anthracycline chemotherapy. | 3 months
determination of radial and circumferential myocardial deformation by echography with 2D strain analysis after 6 months of anthracycline chemotherapy. | 6 months
determination of radial and circumferential myocardial deformation by echography with 2D strain analysis after 9 months of anthracycline chemotherapy. | 9 months
determination of radial and circumferential myocardial deformation by echography with 2D strain analysis after 12 months of anthracycline chemotherapy. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Lafitte, MD-PhD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Service de Cardiologie et Maladies Vasculaires, Hopital du Haut Lévêque, Pessac, France